CLINICAL TRIAL: NCT02117245
Title: Phase I Single Dose Comparative Bioavailability Study Of MGCD265 In Healthy Male And Female Volunteers
Brief Title: Single Dose Comparative Bioavailability Study Of MGCD265 In Healthy Male And Female Volunteers
Status: Completed | Type: Observational
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 265-105
Record Dates: First submitted 2012-05-07; First posted 2014-04-17 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: Food effect on MGCD265 bioavailability in healthy volunteers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pharmacodynamic analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to assess the bioavailability of the MGCD265 formulation following oral administration under fed conditions (Treatment-1) as compared to fasting conditions (Treatment-2) in healthy male and female volunteers.

DETAILED DESCRIPTION:
The study objective is to assess the bioavailability of the MGCD265 formulation following oral administration under fed conditions (Treatment-1) as compared to fasting conditions (Treatment-2) in healthy male and female volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteer
2. Volunteer age of 40 to 65 years
3. Females of childbearing potential using a stable contraceptive method at least 14 days prior to screening and willing to use acceptable birth control methods from 7 days prior to first dose until 30 days after last dose of study drug:
4. Female volunteers will be considered of non childbearing potential and eligible if:

   * Amenorrhea for at least 1 year;
   * Hysterectomy;
   * Bilateral oophorectomy at least 6 weeks prior to first dose;
   * Bilateral tubal ligation at least 6 months prior to first dose;
   * Hysteroscopic sterilization.
5. Male volunteers who agree to be abstinent or use acceptable contraception methods in collaboration with their female partner from the time of taking the first dose until 90 days after the last dose of study drug:

   • Male volunteers who also agree to not donate sperm from the time of taking the first dose until 90 days after the last dose.
6. Volunteer with a body mass index (BMI) greater than or equal to 18.50 and below 30.00 kg/m2
7. Non- or ex smokers for at least 6 months.
8. Availability for the entire study period
9. Motivated volunteer and absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements
10. Clinical laboratory values within the laboratory's stated normal range; or they must be without any clinical significance
11. Have no clinically significant diseases captured in medical history or evidence of clinically significant findings on physical examination and/or clinical laboratory evaluations
12. Willingness to adhere to protocol requirements

The informed consent form must be signed by all volunteers, prior to participation in the study.

Exclusion Criteria:

1. Females who are pregnant or are lactating
2. History of significant hypersensitivity reactions to any substance or drug
3. History or presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with absorption, distribution, metabolism or excretion of drugs
4. Seated blood pressure higher than and equal to 140/90 mmHg at screening
5. Seated blood pressure higher than and equal to 140/90 mmHg before drug administration
6. History or predisposition to cardiovascular illness
7. History or predisposition to thrombotic or hemorrhagic events, bleeding diathesis or coagulopathy, gastrointestinal or other conditions with risk of perforation, presence of a non-healing wound, ulcer or fracture
8. Presence of significant pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
9. No major surgery within 28 days prior to first dose
10. Suicidal tendency, disposition to seizures, state of confusion, clinically relevant psychiatric diseases
11. Presence of out-of-range cardiac interval or ECG abnormalities
12. Maintenance therapy with any drug, or history of drug dependency or alcohol abuse
13. Any clinically significant illness in the previous 28 days before day 1 of study
14. Use of any enzyme-modifying drugs in the previous 28 days before day 1 of study
15. Use of any drugs known to induce or inhibit hepatic metabolism in the previous 28 days before day 1 of study
16. Any history of tuberculosis and/or prophylaxis for tuberculosis
17. Positive urine screening of ethanol and/or drugs of abuse
18. Positive results to HIV, HBsAg or anti-Hepatitis C Virus tests
19. Females who are pregnant
20. Volunteers who took an Investigational Product or donated 50 mL or more of blood in the previous 28 days before day 1 of this study
21. Donation of 500 mL or more of blood in the previous 56 days before day 1 of this study

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy male and female volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Peak Plasma concentration (Cmax) of MGCD265. | 26 days
  Bioavailability of study drug under fed conditions compared to fasting conditions in healthy male and female volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Juretic, Study Director — MethylGene Inc.
Locations (1):
- Algorithme, Laval, Quebec, Canada